CLINICAL TRIAL: NCT01451879
Title: Effects of Immunomodulation Therapy on Anti-rhGAA Immune Response in Subjects With Pompe Disease Receiving rhGAA Enzyme Replacement Therapy
Brief Title: Observational Study for Subjects With Pompe Disease Undergoing Immune Modulation Therapies
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602404; IMN 439-2008 (Other: Legacy study)
Record Dates: First submitted 2011-09-15; First posted 2011-10-14 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Pompe Disease
Keywords: Pompe Disease; Infusion Associated Reaction; Immune-modulation regimen
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Rituximab; miglustat; Morus alba

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood specimens from GAA Ab testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Age 0 months to 65 years: Confirmed diagnosis of Pompe Disease, and clinically prescribed immune modulation regimen with agents such as rituximab, sirolimus, methotrexate, IVIg or other immunomodulatory agents such as pharmacological chaperone Miglustat, N-butyldeoxynojirimycin (NB-DNJ), alone or in combination, at the discretion of their primary/specialist caregiver.
  Interventions: Drug: Rituximab; Drug: Miglustat

INTERVENTIONS:
Drug: Rituximab — Clinically prescribed immune modulation regimen dosage determined by local medical provider.
  Other Names: Rituxan; MabThera; Zytux
Drug: Miglustat — Clinically prescribed immune modulation regimen dosage determined by local medical provider.
  Other Names: Zavesca; N-butyldeoxynojirimaycin; Mulberry extract

SUMMARY:
Hypothesis: the effectiveness of treatment of Pompe Disease with rhGAA enzyme replacement therapy (ERT) is limited at least in part because patients develop antibodies against the provided rhGAA enzyme. Treatment with immunomodulatory drugs may dampen or eliminate the anti-rhGAA immune response in patients receiving ERT, thereby allowing for greater ERT efficacy. Studying the immune response to rhGAA may provide valuable insight into the role of the immune system in the effectiveness of ERT for Pompe Disease.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the effect(s) of medications that alter the immune system on anti-rhGAA immune response in Pompe patients receiving rhGAA enzyme replacement therapy (ERT). The investigators would also like to determine whether treating Pompe Disease with medications that affect the immune system has any effects on the overall health or disease progression of Pompe.

Subjects will be patients between the ages of 0 months and 65 years who have been diagnosed with Pompe Disease, confirmed by mutational analysis and/or GAA enzyme activity assay.

Subjects will be eligible regardless of whether they have begun enzyme replacement therapy prior to enrollment. All Subjects will receive enzyme replacement therapy as standard of care during the course of the Study, although they may not have begun ERT treatment at the time of enrollment. In addition to ERT, subjects may receive an immunomodulatory regimen as part of their standard of care; this may include rituximab, sirolimus, methotrexate, IVIg or other immunomodulatory agents such as pharmacological chaperone N-butyldeoxynojirimycin (NB-DNJ), alone or in combination, at the discretion of their caregiver(s).

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 0 months and 65 years
* diagnosed with early-onset Pompe Disease, confirmed by mutational analysis and/or GAA enzyme assay
* eligible regardless of whether they have begun enzyme replacement therapy prior to enrollment
* all subjects will receive ERT as standard of care during the course of the study, although they may not have begun ERT treatment at the time of enrollment
* subjects may receive an immunomodulatory regimen as part of their standard of care; this may include rituximab, sirolimus, methotrexate, Gamunex, Hizentra, Zavesca or other immunomodulatory agents, alone or in combination, at the discretion of their caregiver(s)

Exclusion Criteria:

* subject is unable to meet the study requirements
* subjects medical condition contraindicates participation or Study Investigators feel that participation is otherwise not in the subject's best interest
* subject does not receive ERT treatment

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of male and female patients age 0-65 years, with a diagnosis of early-onset Pompe Disease. Up to 25 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Anti-rh GAA antibody titers | 52 weeks
  Antibody titer for anti-rh-GAA will be evaluated at baseline and every 4-8 weeks for 52 weeks of participation in the primary study. For subjects who continue participation in the extension study (>52 weeks - 5 years), anti-rh-GAA antibody titers will be evaluated every 12 - 24 weeks.

SECONDARY OUTCOMES:
B-lymphocyte antigen (CD20) level | 52 weeks
  Reports from clinical lab: B-lymphocyte antigen (CD20) will be added to the study record when available every 4-12 weeks during the primary study and every 12 weeks for subjects who participate in the extension study (>52 weeks - 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Byrne, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Elder ME, Nayak S, Collins SW, Lawson LA, Kelley JS, Herzog RW, Modica RF, Lew J, Lawrence RM, Byrne BJ. B-Cell depletion and immunomodulation before initiation of enzyme replacement therapy blocks the immune response to acid alpha-glucosidase in infantile-onset Pompe disease. J Pediatr. 2013 Sep;163(3):847-54.e1. doi: 10.1016/j.jpeds.2013.03.002. Epub 2013 Apr 16. PMID 23601496